CLINICAL TRIAL: NCT00006328
Title: Angiotensin-Converting Enzyme Gene Polymorphism and the Risk of Chronic Allograft Nephropathy
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR00042-1678; M01RR000042 (NIH)
Record Dates: First submitted 2000-10-04; First posted 2000-10-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Kidney Disease
Keywords: Chronic Allograft Nephropathy (CAN); Transplantation immunology; Genetics; Graft Rejection
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Retrospective

SUMMARY:
This study is intended to help doctors learn about the relationships between specific genetic makeup (gene markers) and the development of chronic rejection. This study is being done to see if there is a relationship between genetic patterns and the development of Chronic Allograft Nephropathy (CAN). Medical scientists also hope to learn more about how genetic differences between people determine their response to a drug or a disease by storing a small blood sample in a special "bank". This sample may be tested at some point in the future in an attempt to better understand the factors that may influence rejection, transplantation outcomes and transplant success rates.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be recipients of a renal allograft.
* Study subjects must have evidence of biopsy-proven Chronic Allograft Nephropathy (CAN).
* Control subjects must not have evidence of CAN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Univ. of Michigan Health System, Ann Arbor, Michigan, United States